CLINICAL TRIAL: NCT06978582
Title: Effectiveness and Safety of a Tele-rehabilitation Program Based on Mindful and Conscious Movement-based Exercise vs Conventional Low-intensity Exercise on Fatigue and Related Variables in Patients With Chronic Fatigue Syndrome/ Myalgic Encephalitis (CFS/ME) or Post COVID Syndrome (PCS)
Brief Title: Effectiveness and Safety of a Tele-Rehabilitation Program on Fatigue and Related Variables in Chronic Fatigue Syndrome and Post COVID Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Hermann Fricke Comellas, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0180
Record Dates: First submitted 2025-05-14; First posted 2025-05-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Chronic Fatigue Syndrome/ Myalgic Encephalitis (CFS/ME); Post COVID Syndrome
Keywords: exercise movement techniques; Chronic Fatigue Syndrome; Post COVID Syndrome; mind-body therapies; exercise; pacing; Telerehabilitation
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful and conscious movement-based exercise (Experimental): The intervention will be based on adapted yoga, meditation, breathing exercises, and proprioceptive awareness, in addition to the medical recommendations and pharmacological treatment prescribed by the general practitioner or specialist overseeing each case. The program will last for 12 weeks and will consist of one weekly 45-minute session, with an additional 5 minutes of exercise added each month. Additionally, participants will be encouraged to engage in at least 15 minutes of daily practice with the support of recorded material.
  Interventions: Behavioral: Mindful and conscious movement-based exercise
- Conventional exercise (Active Comparator): The intervention will be based on low-intensity aerobic and strength exercise, in addition to the medical recommendations and prescribed pharmacological treatment provided by the participant's general practitioner or specialist. The program will last for 12 weeks and will consist of one weekly 45-minute session, with an additional 5 minutes of exercise added each month. Additionally, participants will be encouraged to engage in at least 15 minutes of daily practice with the support of recorded material.
  Interventions: Behavioral: Conventional exercise
- Control (No Intervention): The control group will continue with their usual medical care and will not participate in either of the two interventions until all assessments are completed. After the final evaluation, participants in this group will be offered the choice to receive either of the two interventions and will be provided with the corresponding recorded materials.

INTERVENTIONS:
Behavioral: Mindful and conscious movement-based exercise — The program will last for 12 weeks and will consist of one weekly 45-minute session, with an additional 5 minutes of exercise added each month: • 15 minutes of health education. Educational content will focus on self-management, pacing, planning of activity and rest, basic theoretical framework about the conditions, and familiarization with mindful and awareness practices and their purported benefits. • 30 minutes of conscious movement-based exercise practice, increasing by 5 minutes each month and guided by pacing recommendations. Additionally, participants will be encouraged to engage in at least 15 minutes of daily practice with the support of recorded material.
  Arms: Mindful and conscious movement-based exercise
Behavioral: Conventional exercise — The program will last for 12 weeks and will consist of one weekly 45-minute session, with an additional 5 minutes of exercise added each month:
  * 15 minutes of health education. Educational content will now focus on self-management, pacing, planning of activity and rest, basic theoretical framework about the conditions, and the rationale for the impact of exercise in symptom management.
  * 30 minutes of low intensity strength and aerobic exercise practice, with session duration progressively increased by increasing by 5 minutes each month and guided by pacing recommendations.
  Additionally, participants will be encouraged to engage in at least 15 minutes of daily practice with the support of recorded material.
  Arms: Conventional exercise

SUMMARY:
This is a randomized, single-blind clinical trial that aims to evaluate the effectiveness of a tele-rehabilitation program based on mindful and conscious movement-based exercise (including adapted yoga, breathing exercises, and body awareness) compared to conventional exercise (low-intensity strength and aerobic training) and usual medical care (control group) over twelve weeks. The study is for people diagnosed with Chronic Fatigue Syndrome/ Myalgic Encephalitis (CFS/ME) or Post-Covid Syndrome (PCS).

We will also look at how the program affects the autonomic nervous system by measuring heart rate variability (HRV).

All sessions will be delivered remotely via Telehealth, so participants can take part from home. Assessments will be completed online at the beginning of the study, after three months (at the end of the intervention), and again three months later.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of a tele-rehabilitation program based on mindful and conscious movement-based exercise (MBE) in individuals with Chronic Fatigue Syndrome/ Myalgic Encephalitis (CFS/ME) or Post-Covid Syndrome (PCS). The study includes three parallel groups: (1) MBE (including yoga, breathwork, and interoceptive awareness); (2) conventional low-intensity aerobic and strength exercise; and (3) usual medical care as a control. Participants will be randomly assigned to one of the three groups in a 1:1:1 ratio.

All interventions will be delivered via Telehealth, allowing participants to follow the program from home, which increases accessibility and is especially important for people experiencing severe fatigue. The intervention period will last 12 weeks. Both the conscious movement program and the conventional exercise program include a weekly live session of 45 minutes, progressively increased by 5 minutes per month to adapt to tolerance and avoid post-exertional symptom exacerbation. The program is designed with special attention to pacing, allowing participants to self-regulate effort levels based on daily condition and feedback from the body. Participants will also engage in a supportive WhatsApp group and complete digital daily logs.

The primary outcome is fatigue level (measured by the Chalder Fatigue Questionnaire). Secondary outcomes involve heart rate variability (HRV) as an indicator of autonomic function, physical capacity, pain, sleep quality, mental health, interoceptive awareness, quality of life, pain-related fear and somatic vigilance, adverse events, and adherence to the intervention. Assessment points are: baseline (T0), 3 months, at the end of intervention (T1), and follow-up at 6 months (T2). The study follows CONSORT guidelines and is single-blinded (evaluators/statisticians blinded to group assignment).

The expected sample size is 147 participants (49 per group), calculated for sufficient statistical power and accounting for 20% dropout. Recruitment will occur through patient associations, social media, and clinical collaborators. Data analysis will follow an intention-to-treat approach using appropriate mixed models for repeated measures.

The study addresses the need for safe and feasible therapeutic options for people with post-viral fatigue syndromes. It also explores the potential role of interoception and vagal modulation in symptom relief, contributing to a growing body of research on holistic, home-based interventions for chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 and under 70 years of age (to minimize the presence of comorbidities).
* Participants must meet the latest established diagnostic criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and Post-Covid Syndrome, respectively.
* Participants must have access to a computer, tablet, or mobile device with an internet connection to attend videoconference sessions.
* Participants must have a mobile device compatible with the applications Cardiio: Heart Rate Monitor and Welltory, which will be used to measure heart rate (HR) and heart rate variability (HRV), respectively.
* Participants must be able to remain seated in a chair for at least 45 continuous minutes.
* Participants must have fluent comprehension of the Spanish language.
* Any comorbid condition that could explain the symptomatology associated with the syndrome (such as post-infectious organ damage, heart disease, neurological disorders, cancer, severe psychiatric illness, or metabolic syndrome) must have been ruled out by a physician.

Exclusion Criteria:

* Recent suspicion of comorbid conditions that could explain the syndrome's associated symptoms, not yet ruled out by a qualified healthcare professional.
* Inability to use basic software required for participation in the study (e.g., Microsoft Teams, completing a Google Forms questionnaire).
* Unwillingness to make minor adjustments to daily habits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | From baseline to three months after intervention completion
  Fatigue will be measured through the Spanish version of the Chadler Fatigue Scale. It is a 14-item psychometric questionnaire designed to assess the subjective perception of physical and mental fatigue over the past few weeks. Items are rated on a 4-point Likert scale (0 = never, 1 = sometimes, 2 = often, 3 = always). The total score ranges from 0 to 42, with higher scores indicating greater levels of fatigue.

SECONDARY OUTCOMES:
Heart Rate Variability | From baseline to three months after intervention completion
  Welltory Mobile Application (v.4.16.100) is a mobile application that uses photoplethysmography through the phone's camera to measure resting heart rate. Based on these data, it estimates heart rate variability (HRV) parameters, including autonomic balance indicators such as RMSSD and SSDN. The tool has been validated in previous studies for assessing resting HRV, showing a significant correlation with reference medical devices such as electrocardiograms and heart rate monitors (intraclass correlation coefficient > 0.90).
Perceived pain | From baseline to three months after intervention completion
  Perceived pain will be assessed through the Spanish version of the Brief Pain Inventory (BPI), which is a self-administered instrument composed of two sections: pain intensity and the degree of interference in daily activities (such as sleep, mood, work, among others). It consists of 9 items, each rated on a numerical scale from 0 to 10, where higher scores indicate greater pain intensity and/or interference.
Perceived Quality of life | From baseline to three months after intervention completion
  Perceived quality of life will be assessed through the completion of the Spanish version of the SF-36 Health Questionary. It is a widely used tool for measuring health-related quality of life. This instrument consists of 36 items grouped into eight dimensions: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores are transformed to a scale from 0 to 100 for each dimension, with higher scores indicating a better perceived health status in that domain.
Physical function | From baseline to three months after intervention completion
  Physical function will be quantified through the Sit-To-Stand Test. This test is a functional test that measures lower limb muscular endurance. It involves recording the number of repetitions of standing up from and sitting down on a standard armless chair over a 60-second period. The participant must keep their arms crossed over the chest and perform the movement as quickly as possible while maintaining proper technique. This test is a reliable indicator of functional strength and muscular endurance, widely used in both healthy populations and individuals with chronic conditions.
Interoceptive awareness | From baseline to three months after intervention completion
  Interoceptive awareness will be quantified through the Spanish version of the Multidimensional Assessment of Interoceptive Awareness. This is a self-administered 32-item questionnaire that measures interoceptive awareness across eight dimensions, such as attention to internal bodily sensations, emotional regulation through bodily signals, and interoceptive confidence. Each item is rated on a Likert scale from 0 (never) to 5 (always), with higher scores indicating greater interoceptive awareness.
Anxiety and depression levels | From baseline to three months after intervention completion
  Anxiety and depression levels will be measured with the Hospital Anxiety and Depression Scale (HADS) which is a brief questionnaire composed of 14 items divided into two subscales: anxiety (7 items) and depression (7 items). Each item is rated on a scale from 0 to 3, with total scores ranging from 0 to 21 for each subscale. A cutoff score of ≥8 is considered indicative of clinically significant levels of anxiety or depression.
Perceived sleep quality | From baseline to three months after intervention completion
  Perceived sleep quality will be measured with the Pittsburg Sleep Quality Index (PSQI). This is a self-administered questionnaire that assesses sleep quality over the past month. It consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, and the total score ranges from 0 to 21. Scores greater than 5 indicate significant sleep problems.
Fear of movement | From baseline to three months after intervention completion
  Fear of movement will be measured through the Tampa Scale for Kinesiophobia. The Tampa Scale for Kinesiophobia assesses fear of movement related to pain through 17 items rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Total scores range from 17 to 68, with higher scores indicating greater levels of kinesiophobia.
Somatic vigilance | From baseline to three months after intervention completion
  Somatic vigilance will be evaluated using the Anxiety Sensitivity Index (ASI; Spanish version). The ASI consists on 16 items (total score 0-64) assessing fear of anxiety-related bodily sensations, with higher scores denoting greater sensitivity.
Treatment feasibility | From baseline to the end of treatment at 3 months
  Treatment feasibility will be measured through quantification of adherence to treatment and adverse events. An individual digital diary will be used to record this data.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Fricke-Comellas, Principal Investigator, Principal Investigator — University of Seville
Locations (1):
- Facultad de Enfermería, Fisioterapia y Podología. Universidad de Sevilla (Campus Macarena, Perdigones), Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Yes
Only data included in the final study publication will be shared, in accordance with the recommendations of the institutional ethics committee
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be available from the initial protocol registration till the final study publication.
Access Criteria: The information will be available by contacting the principal investigator.

REFERENCES:
- [Background] Fricke-Comellas H, Heredia-Rizo AM, Casuso-Holgado MJ, Salas-Gonzalez J, Fernandez-Seguin LM. Exploring the Effects of Qigong, Tai Chi, and Yoga on Fatigue, Mental Health, and Sleep Quality in Chronic Fatigue and Post-COVID Syndromes: A Systematic Review with Meta-Analysis. Healthcare (Basel). 2024 Oct 11;12(20):2020. doi: 10.3390/healthcare12202020. PMID 39451436
- [Derived] Fricke-Comellas H, Infante-Cano M, Heredia-Rizo AM, Martin-Fernandez A, Escudero-Perez P, Fernandez-Seguin LM. Safety and Effectiveness of an Exercise-Based Telerehabilitation Program in Myalgic Encephalomyelitis and Post COVID Syndrome: Protocol for a Randomized Controlled Clinical Trial. Healthcare (Basel). 2025 Nov 26;13(23):3062. doi: 10.3390/healthcare13233062. PMID 41373279
- See also: Information and contact to participate in the study — https://drive.google.com/drive/folders/1Ge5fJfv5MBSOUL1kSaSC1c_kAUESfZ1F?usp=share_link